CLINICAL TRIAL: NCT02791178
Title: Plaque Evaluation by Optical Coherence Tomography and Its Association With Microvascular Obstruction in Reperfused STEMI Patients - The POMS Study
Brief Title: Optical Coherence Tomography in STEMI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/3034
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from all participants.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- STEMI patients: The patients presenting with a STEMI and undergoing PPCI will be screened and approached to participate in this study.
  All patients to do Optical Coherence Tomography (OCT), Index of Microcirculatory Resistance (IMR) and Cardiac MRI.
  Interventions: Procedure: Optical coherence tomography (OCT); Procedure: Index of microcirculatory resistance (IMR); Other: Cardiac MRI

INTERVENTIONS:
Procedure: Optical coherence tomography (OCT) — Special camera to study part of your heart that was affected
Procedure: Index of microcirculatory resistance (IMR) — Special wire to study part of your heart that was affected
Other: Cardiac MRI — Special scanner if the heart to assess the damage of your heart

SUMMARY:
The overall objective of this research proposal is to use OCT to investigate those morphological culprit plaque characteristics associated with the risk of developing MVO in reperfused STEMI patients.

DETAILED DESCRIPTION:
The specific research objectives include:

1. To use OCT to determine the type of plaque (plaque rupture, plaque erosion or calcified nodule) most associated with the presence and severity of MVO (as measured by IMR and cardiac MRI).
2. To use OCT to investigate the relationship between the extent of tissue protrusion and the amount of residual stent thrombus with the presence and severity of MVO (as measured by IMR and cardiac MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed STEMI as per the in-charge consultant based on presenting history, ECG and angiogram findings.
2. < 12 hours of onset of chest pain.
3. Ability to provide informed consent

Exclusion Criteria:

1. Previous myocardial infarction or coronary artery bypass graft surgery
2. Cardiac arrest or cardiogenic shock
3. Inability to advance the OCT catheter or to obtain good image quality
4. Ostial lesions
5. Significant renal impairment
6. Contraindications for cardiac MRI
7. Contraindication for adenosine (for IMR measurement)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients presenting with a STEMI and undergoing PPCI will be screened and approached to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Derek Hausenloy, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No